CLINICAL TRIAL: NCT00172718
Title: Using 3.3mm Screw Tap to Modify the Standard Implantation Procedure and to Measure the Cutting Resistance for Establishing a More Objective Method to Evaluate the Peri-Implant Bone Quality
Brief Title: Using 3.3mm Screw Tap and Cutting Resistance to Evaluate Bone Quality Around Dental Implant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701264
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2005-02

CONDITIONS: Jaw, Edentulous, Partially; Mouth, Edentulous
MeSH Terms: conditions — Jaw, Edentulous, Partially; Mouth, Edentulous

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Osseointegrated root form implants have been applied successfully in treating fully and partially edentulous patients and patients with single tooth missing. However, the success rate of osseointegrated dental implants was not as good in patients with poor bone quality. The reasons are believed that poor bone quality reduces the initial stability of dental implants and then reduces the success rate. For increasing initial stability of dental implants, some technical modifications are suggested in literature. However, due to lack of an objective method to evaluate bone quality, they are controversial. The purposes of this clinical study are to develop a standard procedure which using cutting resistance measured by Osseocare in surgery to evaluate the bone quality and to compare with the clinical experiences of oral surgeons. The objective outcome, initial stability of dental implant, is measured with Osstell. The analyzed results are also helpful for less experienced surgeons.

DETAILED DESCRIPTION:
Materials & Methods:

1. Patient eligibility: Six implant surgeons will assist the experiment. The subjects are patient who will receive dental implant treatment in Dental department of NTUH. Sixty subjects are offered by six surgeons. They must fully fill the requirements as following

ELIGIBILITY:
Inclusion Criteria:

* No major systemic diseases
* Mouth opening: > 35 mm
* Missing teeth at anterior or premolar area and willing to restored by implantation

Exclusion Criteria:

* Uncomfortable or other condition occurring in the surgical procedure make the measuring unacceptable

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Tong-Mei Wang, DDS, MS, Principal Investigator — National Taiwan University, School of Dentistry; Li-Deh Lin, DDS, PhD, Study Director — National Taiwan University, School of Dentistry
Locations (1):
- Dept. of Dentistry, National Taiwan University Hospital, Taipei, Taiwan